CLINICAL TRIAL: NCT02359708
Title: Recolonisation of Bacteria in Hands and Possible Bacterial Leakage From Glove Cuff in Cardiac Surgery. Differences in Microbial Flora and Recolonisation Between Hospital and Non-hospital Persons. A Controlled Clinical Trial.
Brief Title: Recolonisation of Bacteria in Hands and Possible Bacterial Leakage From Glove Cuff in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Camilla Wistrand, Operating room nurse, Örebro University, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: glovecuff2014
Record Dates: First submitted 2015-01-21; First posted 2015-02-10 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Bacterial Growth
MeSH Terms: interventions — Hand Disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OR nurse group (Experimental): OR nurses (14) who agreed to participate were asked to perform a surgical hand disinfection accordingly to clinic routine. When hands were dry cultures were first obtained at 3 sites, using a moist with saline nylon flocked swab (Copan ESwab, Italia SpA). After hand disinfection; 1) in right hand palm, 2) between index finger and middle finger, 3) nail/cuticle of index finger. When surgery were completed and before disposal of gloves and gown the fourth culture were taken where the glove cuff meets the gown sleeve, under and above, the inner glove of all OR nurses.When gloves were removed cultures were taken again at three sites on the hand, approximately 2-3 hours.
  Interventions: Procedure: Surgical hand disinfection.
- Non-hospital group (Experimental): Non-hospital volunteers who agreed to participate were asked to perform a surgical hand disinfection accordingly to clinic routine. When hands were dry cultures were first obtained at 3 sites, using a moist with saline nylon flocked swab (Copan ESwab, Italia SpA). After hand disinfection; 1) in right hand palm, 2) between index finger and middle finger, 3) nail/cuticle of index finger. This group whore gowns and gloves for approximately 2-3 hours but not kept sterile. The Culture at the glove cuff were left out. When gloves were removed cultures were taken again at three sites on the hand.
  Interventions: Procedure: Surgical hand disinfection.

INTERVENTIONS:
Procedure: Surgical hand disinfection. — Bacterial recolonization

SUMMARY:
This study aims to investigate if recolonisation of the hand flora occur after surgical hand washing and is there a bacterial leakage at the glove cuff site in cardiac surgery? Also investigate if thera are differences in microbial flora and recolonisation between hospital and non-hospital persons.

DETAILED DESCRIPTION:
With emerging antibiotic resistant bacteria it is necessary to try to prevent surgical site infections (SSIs).Not only because of suffering and death but also because of increased costs. For a deep sternal infection the cost can be doubled or even tripled. Sternal wound complications can occur from low numbers up to almost 10%, with different severity, depending on follow up routines In an intraoperative environment causative bacteria often originate from either patient or surgical team. One of many preventing measures is to keep patients and surgical members as sterile as possible when it´s the number of bacteria that overcome the host defense that lead to infection. The most common bacteria causing sternal infection is Coagulase negative staphylococci (CoNS) 46% Staphylococcus aureus, 26% and gram- negative bacteria, 18%. One preventing measure is to wear surgical gloves, and to wear double gloving for easy detection of puncture in outer glove. When using indicator gloves there becomes a dark spot were the hole is which tells you to change the glove. At the glove cuff end it often indicate fluid of some sort by getting dark where the sleeve of the gown meets the glove cuff. One may suspect that the fluid thrives from the hand, and if so does the fluid contains any bacteria from the hands. In open heart surgery surgical team wear their gloves for a long period of time. Research implicates that it occurs some recolonisation of bacteria inside the gloves. Does recolonisation of the hand flora occur after surgical hand washing and is there a bacterial leakage at the glove cuff site? It´s discussed that people that are in contact with hospitals carries more bacteria than others and being admitted to hospital before surgery is a risk factor. It is also known that hospital workers are carriers of more bacteria and possibly also carriers of resistant bacteria. At the other hand hospital workers often wash and disinfect their hands. Are there differences in bacterial recolonization of hand flora between hospital staff at an operating department than people in average society who have little or no contact with hospitals?

ELIGIBILITY:
Inclusion Criteria:

* Operating nurse at the department and non-hospital persons

Exclusion Criteria:

* Participated previously in present study
* Use of gloves with antimicrobial effect
* Patient with a known infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Leakage from gloves at the glove cuff site as bacterial growth cfu/mL | 3 to 4 hours
  Cultures taken after hand wash and after wearing surgical gloves for about 3 hours

SECONDARY OUTCOMES:
Differences between hand flora and its recolonisation, between hospital staff and non-hospital persons showed as bacterial growth, cfu/mL. | 2-3 hours
  Cultures taken after hand wash and after wearing surgical gloves for about 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Wistrand, phd student, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örbro university hospital, Örebro, Sweden

REFERENCES:
- [Derived] Wistrand C, Soderquist B, Falk-Brynhildsen K, Nilsson U. Exploring bacterial growth and recolonization after preoperative hand disinfection and surgery between operating room nurses and non-health care workers: a pilot study. BMC Infect Dis. 2018 Sep 17;18(1):466. doi: 10.1186/s12879-018-3375-3. PMID 30223772